CLINICAL TRIAL: NCT05867472
Title: Advancing Brain Outcomes in Pediatric Critically Ill Patients Sedated With Volatile AnEsthestic Agents: A Pilot Multicentre Randomized Controlled Trial
Brief Title: Advancing Brain Outcomes in Pediatric Critically Ill Patients Sedated With Volatile AnEsthestic Agents
Acronym: ABOVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO - 4285
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Units, Pediatric; Anesthetics, Inhalation; Mechanically Ventilated, Critically Ill Children
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Pilot, multicenter, vanguard randomized controlled trial (RCT) to assess the feasibility of accruing patients, delivering the intervention of inhaled sedatives, and ascertaining outcomes in preparation for a definitive trial to evaluate if inhaled sedatives (intervention) compared to IV agents (comparator) improves delirium (outcome) in mechanically ventilated children (population).
Who Masked: Outcomes Assessor
Masking Description: This is an open label trial that will be blinded to the outcome assessor and data analyst, but not to the clinical team. Blinding is not feasible for the clinical team and patient / family given the easily identifiable differences in the nature of the essential equipment used between the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled sedation - volatile anesthetic (Experimental): The ICU patient will receive Isoflurane. Dosage will be modified as per health care team guidance for the best treatment of the participant.
  Interventions: Drug: Isoflurane Inhalant Product
- IV sedation - standard of care (No Intervention): The ICU patient will receive standard of care, which is IV sedation supplied by the hospital. Dosage will be modified as per health care team guidance for the best treatment of the participant.

INTERVENTIONS:
Drug: Isoflurane Inhalant Product — Isoflurane will be administered using an inhalation device
  Arms: Inhaled sedation - volatile anesthetic

SUMMARY:
The goal of a pilot study is to test a study plan to see if it is appropriate for a larger study. This study plan is looking at whether the use of inhaled sedatives (medications that help people be calm and sleep) can reduce delirium (extreme confusion) in children who need a ventilator (breathing machine) compared to IV or oral sedatives.

The main question[s] it aims to answer are:

* Will people join the study? (recruitment)
* Will participants finish the study?
* Will healthcare teams accept the study procedures?

Participants will be randomized to receive study treatment (inhaled sedation) or standard of care (IV sedation). They will be monitored daily for up to 28 days. They will complete memory, thinking and behaviour tasks after 9-12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients age from 1 month to less than 18 years who need sedation to tolerate mechanical ventilation and will remain ventilated for ≥ 24 hours
2. Receiving IV sedation by infusion or bolus for ≤72h to aid mechanical ventilation (but will be recruited as early as possible)

Exclusion Criteria:

1. Current use of inhaled prostacyclin (high viscosity of prostacyclin impairs vaporizer device) or continuous salbutamol nebulization (impairs gas analyzer function)
2. Family history or personal history of malignant hyperthermia (MH)
3. Allergy to isoflurane, sevoflurane or other volatile inhaled anesthetic gas
4. Metabolic, mitochondrial or myopathy disease e.g., Duchenne muscular dystrophy (volatiles may trigger malignant hyperthermia like reaction)
5. Moribund with expected survival < 24h
6. Known pregnancy or lactation
7. Suspected or evidence of high intracranial pressure (ICP)
8. Not a 'closed ventilator circuit' with potential for gas leak (e.g. uncuffed ETT, bronchopleural fistula, tracheal/trachea-esophageal fistulas, or other sources of "gas leak" from patient circuit that cannot be removed)
9. Prior enrollment in the ABOVE trial

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | 2 years
  Accrual and/or identification of challenges in accruing 60 mechanically ventilated participants (age 1 month to 18 years).

SECONDARY OUTCOMES:
Protocol adherence | 28 days
  The frequency (%) of randomized patients who remain within their designated trial arm and cross-overs. Cross overs may occur from i) drug allergy (rare <0.1%), ii) clinical reason, iii) equipment issues, and iv) health team discomfort using a new intervention.
Attrition | 3 years
  The frequency (%) of randomized patients who are lost to follow up prior to completion of all study outcome measures and the reasons for no follow-up will be documented. Expected loss to follow-up can occur due to i) inter-facility transfers, ii) patient/family withdrawal from the trial, iii) lack of interest in long-term follow-up.
Safety/adverse event rate | From date of consent until the date of resolution or date of death from any cause, whichever came first, assessed up to 13 months
  Adverse events that are assess as related (possibly, probably or definitely) to study intervention, standard of care, or study equipment will be reported. Adverse events that are assess as unrelated to study intervention, standard of care or study equipment will not be reported. Adverse events will be captured from the time of consent until the time of study completion.
Healthcare team satisfaction | Study days 1, 2 & 3
  All health team members (physicians, nurses and respiratory therapists) will be surveyed daily for up to 3 days in both study arms using a 5-point Likert scale satisfaction score. Free text comments will be allowed to better understand barriers and facilitators.

OTHER OUTCOMES:
Feasibility of collecting delirium scores | 28 days
  Proportion of participants who complete delirium (Cornell Assessment of Pediatric Delirium (CAPD)) and coma (Richmond Agitation Sedation Scale (RASS) or COMFORT Behavioural Scale (COMFORT-B)) assessments twice a day.
Delirium-free Coma-free days | 28 days
  The number of full days participants do not experience coma or delirium as assessed by RASS or COMFORT-B for coma and CAPD for delirium.
Anti-psychotic drug use | 28 days
  The administration of anti-psychotic drugs will be captured from baseline until day 28.
Sedative drug use | 28 days
  The administration of sedative drugs will be captured from baseline until day 28.
Blood collection to assess biological markers of delirium, inflammation and brain injury | Study days 1, 2 & 3
  Participants over >2 years old will be able to participate in an optional blood collection sub-study that will look at 60 markers of delirium, inflammation and brain injury.
Feasibility of neurocognitive assessment | 1-year post enrollment
  Proportion of participants who complete 12 month neurocognitive assessment
Neurocognitive scores | 1-year post enrollment
  Assessment of scores from age-appropriate neurocognitive tests completed at 12-months post enrollment
In-hospital mortality | 1 year
  Participant survival status will be captured daily for 28 days and reported at hospital discharge
Ventilator-free days | 28 days
  The use of a ventilator will be captured from baseline until day 28. The number of days a participant does not require a ventilator will be computed.
ICU-free days | 28 days
  ICU discharge date will be captured and compared to admission date to determine number of days the participant was not in the ICU up to 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jerath, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital - London Health Sciences Centre, London, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario